CLINICAL TRIAL: NCT00504257
Title: A Phase II Trial of Avastin in Combination With Docetaxel in Patients With Recurrence of Epithelial Carcinoma of the Ovary/Fallopian Tube/Peritoneum Within 12 Months of Platinum Therapy
Brief Title: Avastin in Combination With Docetaxel in Ovarian/Fallopian Tube/Peritoneum Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14920; AVF3823s (Other: Genentech); IST13070 (Other: Sanofi-Aventis US Inc.)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Malignant Tumor of Peritoneum
Keywords: recurrent ovarian epithelial cancer; recurrent primary peritoneal cavity cancer; recurrent fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin and Docetaxel (Experimental): Combination Therapy: Immunotherapy (Avastin) and Chemotherapy (Docetaxel) as outlined in Intervention descriptions. Avastin: 15 mg/kg, In 100 ml normal saline (NS) IV infusion over 90 +/- 15 minutes, Day 1, every 21 day cycle. Docetaxel: 40 mg/m^2, In 250 ml 5% dextrose in pure water (D5W) or NS IV infusion over 1 hour in a non-pvc container and through a polyethylene-lined set, Day 1, 8, every 21 day cycle. Response assessment every 3 cycles (9 weeks).
  Interventions: Drug: Avastin; Drug: Docetaxel

INTERVENTIONS:
Drug: Avastin — Day 1, every 21 day cycle
  Other Names: Avastin™; bevacizumab
Drug: Docetaxel — Day 1, 8, every 21 day cycle
  Other Names: TAXOTERE®

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the combination of Avastin and Docetaxel in the treatment of women with platinum sensitive recurrent epithelial ovarian cancer within 12 months of platinum chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Pathologically confirmed epithelial ovarian cancer, peritoneal serous cancer, or fallopian tube cancer
* Patient's disease recurrence or progression occurs between 0 to 12 months (1 to 365 days) from prior platinum-containing chemotherapy regimen. Patients, however, may not receive study drug until at least 28 days from prior chemotherapy.
* The patient may have received up to three prior chemotherapy regimens for the treatment of this malignancy. Patients who may have received prior treatment with paclitaxel and/or a platinum compound will be allowed. Rechallenge with the same platinum based regimen is considered 1 prior regimen. Patients who have been treated with consolidation treatment are allowed and the consolidation will not be considered a separate regimen. Hormonal therapy (i.e. progesterones, estrogens, anti-estrogens, aromatase inhibitors) will not be considered a prior chemotherapy regimen.
* Measurable or evaluable disease either by the Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST) or cancer antigen (CA)125 criteria [Journal of the National Cancer Institute (JNCI), Vol. 96, No. 6, March 17, 2004, Vergote JNCI 2000]
* At least 4 weeks since major surgery, with full recovery
* At least 3 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside of the radiation port.
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2
* Hematologic (minimal values): Absolute neutrophil count >/= 1,500/mm^3, Hemoglobin >/= 8.0 g/dL (transfusions allowed), Platelet count >/= 100,000/mm^3
* Hepatic: Total Bilirubin </= upper limit of normal (ULN), alanine transaminase (AST) and alanine transaminase (ALT) and alkaline phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the 2 values (AST or ALT) should be used.
* Women of childbearing potential must have a negative pregnancy test.
* Patients of childbearing potential must be willing to consent to using effective contraception while on treatment and for 3 months following the completion of treatment.

Exclusion Criteria:

Prior treatment with Docetaxel or Avastin

* Concurrent immunotherapy or hormonal therapy for the specific purpose of treatment for the ovarian cancer. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to enrollment in order for the patient to be eligible to participate in this trial. Continuation of hormonal replacement therapy is allowed.
* Peripheral neuropathy >/= grade 2
* History of a severe hypersensitivity reaction to Docetaxel, Avastin, or to other drugs formulated with polysorbate (Tween) 80.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study of Avastin
* Blood pressure of >150/100 mmHg Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months prior to Day 1
* History of stroke within 6 months prior to Day 1
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein: creatinine ratio >/= 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Evidence of malignancy in the last 5 years, other than nonmelanoma cutaneous carcinomas
* History of hemoptysis (bright red blood of 1/2 teaspoon or more) within last 3 months
* Patients believed to possibly be at higher than average risk of perforation will be excluded from study. This includes symptoms or findings of partial or complete bowel obstruction, history of fistula, patients requiring parenteral nutrition and hydration, and those with history of prior perforation due to tumor or perforation within last 6 months from other causes.
* Inability to comply with study and/or follow-up procedures.
* Patients who are not on a stable dose of anticoagulation therapy. Patients who are on a stable anticoagulation regimen, including coumadin or low molecular-weight heparin, will not be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Wenham, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (4):
- United States (4):
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Duke Cancer Institute, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2007 and February 2011, 45 patients were screened.
Period: Overall Study
Arm/Group | Avastin and Docetaxel
Started | 45
Completed | 41
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — ineligible histology | 2

BASELINE CHARACTERISTICS:
Population: Participants who were evaluable for the outcome measures.
Arm/Group | Avastin and Docetaxel
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 58.2 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Six Month Progression Free Survival (PFS)
Description: Percentage of participants with PFS at six months. PFS: Period from study entry until disease progression, death due to disease progression, or date of last contact.
  Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, progression of non-target lesions, or the appearance of one or more new lesions.
Time Frame: 6 months per participant
Population: All evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin and Docetaxel
Number analyzed (Participants) | 41
percentage of participants | 43.9 [28.6 to 58.2]

2. Secondary Outcome: Median Progression Free Survival
Description: PFS: Period from study entry until disease progression, death due to disease progression, or date of last contact.
  Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, progression of non-target lesions, or the appearance of one or more new lesions.
Time Frame: Up to 5 years
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avastin and Docetaxel
Number analyzed (Participants) | 41
months | 5.2 [4.4 to 7.2]

3. Secondary Outcome: Overall Response Rate (RR)
Description: Overall Response: Complete Response (CR) + Partial Response (PR). To determine the response rate (RR) of the investigational treatment regimen. Response and progression were evaluated in the study by using the Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST) method or modified Rustin Criteria for CA-125 measurements.
Time Frame: Up to 5 years
Population: Response Rate (RR) evaluable patients included all patients who received at least 2 cycles of treatment and at least one tumor assessment or had demonstrated clinical progression.
Measure: Number; unit: participants
Arm/Group | Avastin and Docetaxel
Number analyzed (Participants) | 38
participants | 22

4. Secondary Outcome: Occurrence of Grade 3 or 4 Toxicity
Description: Number of participants with Grade 3 or 4 Toxicity based on 278 treatment cycles. Toxicity was graded per the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Up to 4 years
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | Avastin and Docetaxel
Number analyzed (Participants) | 41
participants | 27

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS): defined as observed length of life from entry onto the protocol to death, or for living patients, date of last contact (regardless of whether or not this contact is on a subsequent protocol). Survival (PFS and OS) were analyzed using the Kaplan-Meier method with standard errors based on Greenwood's formula.
Time Frame: Up to 5 years
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avastin and Docetaxel
Number analyzed (Participants) | 41
months | 12.4 [10.0 to 21.9]

ADVERSE EVENTS:
Time Frame: 4 years
Description: Participants who received 1 to 278 treatment cycles.
Arm/Group | Avastin and Docetaxel
Serious Adverse Events (participants affected / at risk) | 27/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin and Docetaxel (N=41)
Fistula, GI - Colon/cecum/appendix (Gastrointestinal disorders) | 1
Obstruction, GI - Small bowel, NOS (Gastrointestinal disorders) | 3
Perforation, GI - Small bowell, NOS (Gastrointestinal disorders) | 2
Febrile neutropenia (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Pain - Back (General disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6
Fatigue (asthemia, lethargy, malaise) (General disorders) | 5
Anorexia (Gastrointestinal disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1
Pain - Stomach (General disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 1
Pain - Kidney (General disorders) | 1
Neuropathy: sensory (Musculoskeletal and connective tissue disorders) | 2
Platelets (Blood and lymphatic system disorders) | 1
Ileus, GI (functional obsturction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin and Docetaxel (N=41)
Diarrhea (Gastrointestinal disorders) | 19
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 16
Anorexia (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 15
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 12
Gastrointestinal - other (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 8
Heartburn/dyspepsia (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Distention/bloating, abdominal (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 5
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 18
Constitutional Symptoms - Other (General disorders) | 10
Insomnia (General disorders) | 5
Rigors/chills (General disorders) | 4
Weight gain (General disorders) | 4
Weight loss (General disorders) | 4
Fever (in the absence of neutropenia) (General disorders) | 3
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 25
Nail changes (Skin and subcutaneous tissue disorders) | 18
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pain - abdomen, NOS (General disorders) | 13
Pain - Head/headache (General disorders) | 7
Pain - Other (General disorders) | 7
Pain - Oral cavity (General disorders) | 5
Pain - Back (General disorders) | 3
Pain - Chest/thorax, NOS (General disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 12
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 17
Dizziness (General disorders) | 5
Neuropathy: motor (Nervous system disorders) | 3
Watery eye (epiphora, tearing) (Eye disorders) | 24
Vision-blurred vision (Eye disorders) | 4
Dry eye syndrome (Eye disorders) | 3
Ocular/Visual - Other (Eye disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 12
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 9
Lymphopenia (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 6
Hemorrhage, pulmonary/upper respiratory - Nose (General disorders) | 16
Hemorrhage/Bleeding - Other (General disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3
Febrile neutropenia (fever of unknown origin) (Infections and infestations) | 3
Infection with unknown ANC - Urinary tract, NOS (Infections and infestations) | 3
Allergic rhinitis (Immune system disorders) | 7
Hot flashes/flushes (Endocrine disorders) | 9
Hypertension (Cardiac disorders) | 6
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 4
Edema: limb (Blood and lymphatic system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes